CLINICAL TRIAL: NCT04446221
Title: Long Term Follow-Up of Post Neck Pain Patients Accompanying Ossification of Posterior Longitudinal Ligament Treated With Integrated Complementary and Alternative Medicine: Observational Study
Status: Completed | Type: Observational
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Other Study IDs: JS-CT-2020-05
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: OPLL; Medicine, Korean Traditional
Keywords: acupuncture therapy; herbal medicine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: phone survey — A questionnaire about the current symptoms and satisfaction for received treatment will be conducted over the phone for patients.

SUMMARY:
The purpose of this study is to reveal the effectiveness and safety of integrative Korean medicine for Ossification of Posterior Longitudinal Ligament(OPLL) by observation inpatients treated with integrative Korean medicine.

This study is a prospective observational study. The subjects for study are patients diagnosed with OPLL and who have been admitted to four Jaseng Hospital of Korean medicine (Gangnam, Bucheon, Daejeon, and Haeundae) for 2016.04.01-2019.12.31.

Medical records of selected patients will be analyzed, and telephone surveys will be conducted for each patient. The survey questions are Numeric ratinc scale (NRS), Vernon-Mior Neck Disability Index (NDI), quality of life, and Patient Global Impression of Change (PGIC), etc.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with OPLL by C spine X-ray or MRI or CT
* Paithents who was admitted to Jaseng hospital of Korean medicien.
* Patients have agreed to participate the study.

Exclusion Criteria:

* Patient hospitalized under 3 days
* Patients who have been diagnosed with certain serious diseases that may cause disturbance to interpretation of conclusion (cardiovascular problems, kidney disease, diabetic neuropathy, dementia, epilepsy, and so on)
* Patients who have been diagnosed with certain serious diseases that may cause back pain or neck pain (tumor metastases to the spine, fibromyalgia, rheumatoid arthritis, gout, and so on)
* Patients had cervical spinal surgery within 3 months
* Patients diagnosed with C spine fracture by C spine X-ray or MRI or CT
* Patients deemed unable to participate in the clinical research by other researchers
* Patients haven't agreed to participate the study.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The subjects for study are patients diagnosed with OPLL and who have been admitted to four Jaseng Hospital of Korean medicine (Gangnam, Bucheon, Daejeon, and Haeundae) for 2016.04.01-2019.12.31
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) | Finish survey by September 2020
  NRS uses an 11-point scale to evaluate current neck pain and radiating pain where no pain is indicated by '0', and the worst pain imaginable by '10'. NRS was assessed at admission, 2 weeks after admission, discharge, and long term follow up.

SECONDARY OUTCOMES:
Vernon-Mior Neck Disability Index (NDI) | Finish survey by September 2020
  NDI is a 10-item questionnaire developed to evaluate the degree of disability for neck back pain. Each item is divided into 6 levels, and 0 to 5 points are awarded. The higher the score, the greater the degree of disability. We will conduct an validated Korean NDI questionnaire
The five level version of EuroQol-5 Dimension (EQ-5D) | Finish survey by September 2020
  EQ-5D is most widely used as a method of indirectly calculating the quality of life from various aspects. The EQ-5D-5L consists of 5 questions (mobility, self-care, usual activities, pain, anxiety/depression) that ask about the current state of health, and answers each question with 5 likert. (1=I have no problems about, 2=I have slight problems about, 3=I have moderate problems about, 4=I have severe problems about, 5=I am unable to about) In this study, the validated Korean version questionnaire will be used.
Patient Global Impression of Change (PGIC) | Finish survey by September 2020
  PGIC is an indicator that evaluates the improvement of patients in 7 steps, and the subject responds with improvement of functional limitation after treatment with 7 likert. (1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse).
Spine surgery | Finish survey by September 2020
  The number of spinal surgery after discharge
Current symptoms survey | Finish survey by September 2020
  Pain, neurological problems, etc.
Treatment after discharge survey | Finish survey by September 2020
  Treatment history in the last 3 month
Satisfaction with integrative Korean medicine survey | Finish survey by September 2020
  Preference for integrative Korean medicine, satisfaction with integrative Korean medicine, How helpful hospitalization has been for returning to work and adjusting to daily life.

CONTACTS AND LOCATIONS:
Locations (1):
- Jaseng Medical Foundation, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No